CLINICAL TRIAL: NCT01747174
Title: Randomized Controlled Trial Comparing Intracoronary Administration of Adenosine or Sodium Nitroprusside to Control for Attenuation of Microvascular Obstruction During Primary Percutaneous Coronary Intervention
Brief Title: REperfusion Facilitated by LOcal Adjunctive Therapy in ST-elevation Myocardial Infarction
Acronym: REFLO-STEMI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CLRN 53469; 2010-023211-34 (EudraCT Number); 09/150/28 (Other Grant/Funding Number: NIHR EME)
Record Dates: First submitted 2012-11-20; First posted 2012-12-11 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: ST-elevation Myocardial Infarction (STEMI)
Keywords: STEMI; Microvascular Obstruction; No-reflow; Adenosine; Sodium Nitroprusside
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Nitroprusside

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Std PCI + Intra-coronary (IC) Adenosine (Experimental): IC Adenosine in to IRA (following thrombus aspiration) with further dose via guide catheter following coronary stent deployment.
  Interventions: Drug: IC Adenosine; Procedure: Standard PCI
- Std PCI + IC Sodium Nitroprusside (SNP) (Experimental): IC SNP in to IRA (following thrombus aspiration) with further dose via guide catheter following coronary stent deployment.
  Interventions: Drug: IC Sodium nitroprusside (SNP); Procedure: Standard PCI
- Std PCI (Active Comparator): Standard PCI only
  Interventions: Procedure: Standard PCI

INTERVENTIONS:
Drug: IC Adenosine — IC Adenosine 1mg injected distally via micro-catheter in to IRA following thrombus aspiration with further dose (1mg if IRA is RCA otherwise 2mg) via guide catheter following coronary stent deployment.
  Other Names: Adenocor
  Arms: Std PCI + Intra-coronary (IC) Adenosine
Drug: IC Sodium nitroprusside (SNP) — IC SNP 250mcg injected distally via micro-catheter distally in to IRA following thrombus aspiration with further 250 mcg dose delivered via guide catheter following coronary stent deployment.
  Other Names: Sodium pentacyanonitrosylferrate(II); Sodium nitroferricyanide; Sodium pentacyanonitrosylferrate; SNP
  Arms: Std PCI + IC Sodium Nitroprusside (SNP)
Procedure: Standard PCI — PCI procedure with thrombectomy (via aspiration catheter) and bivalirudin given as standard.

SUMMARY:
The purpose of this study is to determine whether intra-coronary adenosine or sodium nitroprusside (SNP) delivered selectively via a thrombus aspiration catheter (or if unsuccessful via a coronary microcatheter) following thrombus aspiration in Primary Percutaneous Coronary Intervention (P-PCI) reduces microvascular obstruction (MVO) parameters and infarct size as measured with cardiac MRI, compared with standard treatment following thrombus aspiration in patients presenting with ST-elevation myocardial infarction (STEMI).

DETAILED DESCRIPTION:
>100,000 patients suffering STEMI present in the UK each year. P-PCI in the UK is increasing exponentially. In 2004 there were <1500 P-PCI and in 2007 and 2008 these figures had increased to 5902 and 9224 respectively (BCIS database).

Although P-PCI delivered quickly is more effective than thrombolysis, the efficacy of this, essentially mechanical, technique is limited by the unpredictable phenomenon of no-reflow and the under-stated lesser degrees of MVO. As more UK centres adopt P-PCI the dilemma of how to attenuate MVO will remain. Currently there is no consensus on the optimal management to prevent or attenuate MVO particularly when thrombus laden lesions are treated with P-PCI.

There is divergent clinical practice, even within institutions, in the UK and worldwide. This is because there is no solid evidence base to inform clinicians. The current options for interventional cardiologists are:

1. Routinely aspirate thrombus and give IC vasodilator during the intervention but only in high burden thrombus formation lesions.
2. Perform a standard P-PCI only and then give IV vasodilator if angiographic no-reflow develops.
3. Routinely consider that angiographically silent MVO (i.e a grade below true "no-reflow") may have important impact on infarct size and clinical outcome and treat prophylactically.

Few if any clinicians follow this thinking. Indeed, it appears impossible to predict the incidence of (no-reflow/MVO) from the presenting angiogram (pre- or post- wire or balloon) and it can be argued that irrespective of thrombus burden it would be better to undertake prophylactic treatment in all patients, following the use of aspiration catheter, with delivery of agents able, in theory at least, to reduce (angiographically undetectable) MVO. Several studies of IC adenosine or SNP have shown favourable effects in attenuating MVO. However, the size of effect with either drug and whether indeed there is a difference between them in reducing MVO and infarct size is undetermined.

The objectives of our proposed study are to determine:

1. Whether adjunctive pharmaco-therapy at time of P-PCI and following thrombus aspiration, reduces CMR-determined MVO and infarct size.
2. Whether there is a difference between adenosine and SNP in reducing CMR-detected MVO and infarct size, both given selectively and distally via a thrombus aspiration catheter or a coronary microcatheter.
3. The correlation of angiographic, including the recently designed computer-assisted myocardial blush quantification 'Quantitative Blush Evaluator'(QuBE), and other myocardial perfusion markers, with CMR detected MVO and infarct size, as well as with clinical outcome (MACE) at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years age.
* Informed ASSENT (verbal consent) prior to angiography.
* STEMI ≤ 6 hrs of symptom onset, requiring primary reperfusion by PCI.
* Single-vessel coronary artery disease (non culprit disease ≤70% stenosis at angiography)
* TIMI flow 0/I at angiography.

Exclusion Criteria:

* Contraindications to: P-PCI *, CMR**, contrast agents, or study medications: Adenosine***, SNP****, Aspirin, Thienopyridine and Bivalirudin.
* SBP ≤ 90mmHg
* Cardiogenic Shock
* Previous Q wave myocardial infarction
* Culprit lesion not identified or located in a by-pass graft
* Stent thrombosis.
* Left main disease.
* Known severe asthma.
* Known stage 4 or 5 chronic kidney disease (eGFR<30ml/min).
* Pregnancy.

Notes:

* * Exclusion criteria for P-PCI (presentation timing, inadequate arterial access etc); patient unable to tolerate "prolonged" PCI procedure (in operators' opinion).
* ** Absolute contra-indication to CMR (Pacemaker, ICD, intra-cranial metal clips).
* *** Contraindications to Adenosine (known hypersensitivity to Adenosine, sick sinus syndrome, second or third degree atrio-ventricular block - except in patients with functioning artificial pacemaker, long QT syndrome has been defined as QTc > 450 ms at baseline). ECG will be undertaken just after the first dose of the study drug and QT/QTc will be recorded and compared to the baseline. If the QTc recorded after the first dose of the study drug exceeds 450ms or there is an increase in the QT/QTc of > 60 ms from baseline, the second dose will be abandoned and this will be recorded.
* **** Contraindications to SNP (known hypersensitivity to SNP, compensatory hypertension - as may be seen in arteriovenous shunts or coarctation of the aorta, high output failure, congenital optic atrophy or tobacco amblyopia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2011-10; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
CMR measured infarct size (% LV mass) | 48-72 hours post procedure

SECONDARY OUTCOMES:
CMR incidence and extent of MVO (% LV mass) | 48-72 hours post procedure
CMR measured myocardial salvage index, haemorrhage, LV EF and volumes | 48-72 hours post procedure
Myocardial Blush Grade assessed by validated computer software 'Quantitative Blush Evaluator' (QuBE | During P-PCI
Incidence pre- and post- procedure angiographic true "no-reflow" | During P-PCI
Any in-patient clinical events | Within 6 months from presentation with, and PCI for, STEMI
  Includes: coronary artery re-occlusion, need for repeat PCI, recurrent chest pain with new ECG changes, incidence of clinical heart failure (symptoms plus basal crackles plus X-ray evidence of pulmonary congestion) and proven cerebrovascular accident (CVA).
Overall MACE | 1 month
  MACE: composite of death, need for target lesion revascularization, recurrent MI, severe heart failure, and CVA.
Degree of ST segment resolution on ECG | Assessed immediately following P-PCI (expected on average 1 hour)
Echocardiographic assessment of LV | 6-8 weeks post-procedure/MI
  To include end systolic/diastolic volumes, EF +/- wall motion index
Corrected TIMI Frame Count | During procedure
  TIMI frame count or TFC is defined as the number of cineframes required for contrast to reach a standardized distal coronary landmark in the culprit vessel.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony H Gershlick, MBBS, FRCP, Principal Investigator — University of Leicester
Locations (4):
- United Kingdom (4):
  - Glenfield Hospital, Leicester, Leicestershire
  - Freeman Hospital, Newcastle upon Tyne, Tyne and Wear
  - University Hospital, Coventry, West Midlands
  - Leeds General Infirmary, Leeds, West Yorkshire

REFERENCES:
- [Derived] Nazir SA, McCann GP, Greenwood JP, Kunadian V, Khan JN, Mahmoud IZ, Blackman DJ, Been M, Abrams KR, Shipley L, Wilcox R, Adgey AA, Gershlick AH. Strategies to attenuate micro-vascular obstruction during P-PCI: the randomized reperfusion facilitated by local adjunctive therapy in ST-elevation myocardial infarction trial. Eur Heart J. 2016 Jun 21;37(24):1910-9. doi: 10.1093/eurheartj/ehw136. Epub 2016 May 4. PMID 27147610
- [Derived] Nazir SA, Khan JN, Mahmoud IZ, Greenwood JP, Blackman DJ, Kunadian V, Been M, Abrams KR, Wilcox R, Adgey AA, McCann GP, Gershlick AH. The REFLO-STEMI trial comparing intracoronary adenosine, sodium nitroprusside and standard therapy for the attenuation of infarct size and microvascular obstruction during primary percutaneous coronary intervention: study protocol for a randomised controlled trial. Trials. 2014 Sep 25;15:371. doi: 10.1186/1745-6215-15-371. PMID 25252600